CLINICAL TRIAL: NCT00172003
Title: Effect of Zoledronic Acid in Patients With Renal Cell Cancer and Bone Metastasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EDE15
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Renal Cell Cancer; Neoplasm Metastasis
Keywords: Renal Cell Cancer; Bone metastasis; Skeletal related event; Renal Cell Cancer patients with bone metastasis
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronic acid (Experimental): Zoledronic acid, dosage according to calculated creatinine clearance, administered as a 15 minute infusion every 3 weeks for 12 months. Study infusion visits should occur not earlier than the scheduled visit and no later than 3 days after the scheduled visit. The dose of zoledronic acid in patients with baseline creatinine clearance > 60 mL/min was recommended to be 4 mg infused over no less than 15 minutes.
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
It is the aim of this clinical study to evaluate the skeletal-related event rate under therapy with zoledronic acid in patients with renal cell cancer having at least one cancer-related bone lesion.

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed diagnosis of renal cell carcinoma with none, one or, at maximum, 2 of the following risk factors:

  1. Karnofsky performance status less than 80%
  2. Lactate dehydrogenase greater than 1.5 times upper limit of normal
  3. Hemoglobin less than lower limit of normal
  4. Absence of nephrectomy
* Patients must have evidence of at least one cancer-related bone lesion. If diagnosis of bone metastases in bone scan or magnetic resonance imaging (MRI)-QuickScan is unclear radiographic (X-ray, computed tomography [CT] or MRI) confirmation of at least one focus is required.
* ECOG performance status of 0, 1 or 2.
* Life expectancy of ≥ 6 months
* Adequate liver function - serum total bilirubin concentration less than 1.5 x upper limit of normal value
* Patient has given written informed consent prior to any study-specific procedures

Exclusion Criteria:

* Only patients who received 3 or less applications of an i.v. Bisphosphonate in the past are eligible
* Previous radiation therapy to bone (including therapeutic radioisotopes such as strontium 89) is allowed. However, other loci of bone metastasis must be present, which were not treated with radiation therapy and thus can be assessed for primary and secondary endpoints.
* Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute. Creatinine clearance (CrCl) is calculated using the Cockcroft-Gault formula: CrCl = [140-age (years)] x weight (kg) {x 0.85 for female patients} [72 x serum creatinine (mg/dL)]
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or ≥ 12.0 mg/dl (3.00 mmol/L)
* Patients with clinically symptomatic brain metastases
* History of diseases with influence on bone metabolism such as Paget's disease and primary hyperparathyroidism
* Severe physical or psychological concomitant diseases that might impair compliance with the provisions of the study protocol or that might impair the assessment of drug or patient safety, e.g. clinically significant ascites, cardiac failure, NYHA III or IV, clinically relevant pathologic findings in ECG.
* Known hypersensitivity to Zometa® (zoledronic acid) or other bisphosphonates
* Pregnancy and lactation
* Women of childbearing potential not on a medically recognized form of contraception (i.e., oral contraceptives or implants, intrauterine device [IUD], vaginal diaphragm or sponge, or condom with spermicide)
* Use of other investigational drugs (drugs not marketed for any indication) within 30 days prior to the date of study inclusion
* Use of other investigational drugs (drugs not marketed for any indication) within 30 days prior to the date of study inclusion
* Participation in another trial
* Known history or present abuse of alcohol or drugs (accepted social alcohol usage will not exclude the patient)
* Subjects who, in the opinion of the investigator, are unlikely to cooperate fully during the study
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Rate of skeletal complications | continuous

SECONDARY OUTCOMES:
Time to first skeletal complication | from first application of Zometa until confirmed skeletal related event (SRE)
Bone pain | every 9 weeks
Time to overall progression of disease | continuous
Overall survival | continuous
Bone turnover parameters | every 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis investigative Site, Offenbach, Germany

REFERENCES:
- [Result] Tunn UW, Stenzl A, Schultze-Seemann W, Strauss A, Kindler M, Miller K, Wirth MP, Zantl N, Schulze M, May C, Ruebel A, Birkholz K, Gruenwald V. Positive effects of zoledronate on skeletal-related events in patients with renal cell cancer and bone metastases. Can J Urol. 2012 Jun;19(3):6261-7. PMID 22704310